CLINICAL TRIAL: NCT04891913
Title: Phase Ib Clinical Study to Evaluate Safety, Tolerance，Pharmacokinetics and Efficacy of SY-007 After Intravenous Injection in Acute Ischemic Stroke Subjects
Brief Title: SY007 in Patients With Acute Ischemic Stroke
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided to suspend the process
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SY007002
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15mg SY-007/ Placebo Repeat Dose (Experimental): Intravenous infusion of 15mg SY-007 or placebo twice a day for seven consecutive days.
  Interventions: Drug: SY-007/ Placebo 15mg
- 30mg SY-007/ Placebo Repeat Dose (Experimental): Intravenous infusion of 30mg SY-007 or placebo twice a day for seven consecutive days.
  Interventions: Drug: SY-007/ Placebo 30mg
- 60mg SY-007/ Placebo Repeat Dose (Experimental): Intravenous infusion of 60mg SY-007 or placebo twice a day for seven consecutive days.
  Interventions: Drug: SY-007/ Placebo 60mg

INTERVENTIONS:
Drug: SY-007/ Placebo 15mg — 15 mg SY-007/ Placebo, the dosing interval is 12 hours ±2 hours for 7 consecutive days.
  Arms: 15mg SY-007/ Placebo Repeat Dose
Drug: SY-007/ Placebo 30mg — 30 mg SY-007/ Placebo, the dosing interval is 12 hours ±2 hours for 7 consecutive days.
  Arms: 30mg SY-007/ Placebo Repeat Dose
Drug: SY-007/ Placebo 60mg — 60 mg SY-007/ Placebo, the dosing interval is 12 hours ±2 hours for 7 consecutive days.
  Arms: 60mg SY-007/ Placebo Repeat Dose

SUMMARY:
This Phase 1b multiple center, randomized, double-blind, placebo-controlled study is a dose escalation trial evaluating the safety, tolerability, PK characteristics and efficacy of SY-007 after injection in acute ischemicstroke patients. The immunogenicity of SY-007 will be evaluated and this study will provide the recommended dosage for subsequent clinical trials.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged from18 Years to 80 Years
* Within 24h after the onset of stroke symptoms (time the patient was last seen well)
* Score range from 4 to 20 points, inclusive, on the NIHSS at randomization
* Prior to index stroke, patient was able to perform basic activities of daily living without assistance, mRS score≤1
* Absence of intracranial hemorrhage on brain CT or MRI
* Patients or legal representatives can give informed consent

Key Exclusion Criteria:

* Venous thrombolytic therapy or endovascular treatments have been applied for patients; or Patients plan to conduct these kind of treatments.
* Glasgow score of Patients ≤8
* Patients are receiving oral anticoagulants or INR>3.0
* Baseline blood platelet counts <80*109/L
* NIHSS score could not been obtained at baseline
* FPG levels < 50mg/dL or >400mg/dL
* Patients with Kidney disorder eGFR <30 mL/min or patients need dialysis
* Patients with Acute and Chronic hepatitis, or Liver diseases (AST or/and ALT >2 × ULN(upper limit normal))
* systolic blood pressure≥220mmHg or/and diastolic blood pressure≥120mmHg ; or Blood pressure under 90/60mmHg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance of SY-007 | From Day 0 to Day 90
  Number of patients with treatment-emergent adverse events and number of patients who died over 90 days

SECONDARY OUTCOMES:
Pharmacokinetics of SY-007 | From Day 0 to Day 7
  Peak Plasma Concentration (Cmax)
Pharmacokinetics of SY-007 | From Day 0 to Day 7
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics of SY-007 | From Day 0 to Day 7
  Time to Cmax (Tmax)
Pharmacokinetics of SY-007 | From Day 0 to Day 7
  Terminal half life (T½)
Pharmacokinetics of SY-007 | From Day 0 to Day 7
  Clearance (CL)
Pharmacokinetics of SY-007 | From Day 0 to Day 7
  Volume of distribution
Percentage of Participants With Excellent Outcome in Modified Rankin Scale（mRS) Score at Day 8, Day30, Day60, Day90 | Day 8, Day30, Day60, Day90
  Excellent mRS is defined as mRS score of 0 or 1
Modified Rankin Scale Score at Day 8, Day30, Day60, Day90 | Day 8, Day30, Day60, Day90
  Modified Rankin Scale Score range from 0 to 5，higher score mean a worse outcome.
Percentage of Participants With National Institute of Health Stroke Scale (NIHSS) range from 0 to 1 at Day 8, Day30 | Day 8, Day30
Change From Baseline in NIHSS Score at Day 8, Day30 range from 0 to 1 at Day 8, Day30 | Day 8, Day30
Percentage of Participants With Excellent Outcome in Barthel index (BI) Score at Day 8, Day30, Day60, Day 90 | Day 8, Day30, Day60, Day 90
  Excellent BI outcome is defined as a score of >=95. BI consists of 10 items that measure a participant's daily functioning, specifically the activities of daily living and mobility.
Change of Cerebral infarction volume before and after treatment | Baseline, Day 8, Day30
Immunogenicity of SY-007 | From Day 0 to Day 30
  Anti-Drug antibody evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, China